CLINICAL TRIAL: NCT04179227
Title: Developing a Social Media-Delivered Intervention
Brief Title: Focus Group in Collecting Feedbacks From Indoor Tanning Bed Users for Social Media-Delivered Intervention Development
Status: Terminated | Type: Observational
Why Stopped: PI left institution.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Professor and Associate Director of Population Science, Rutgers Cancer Institute of New Jersey
Other Study IDs: Pro20170000136; NCI-2018-00058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20170000136; 131703 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Health Status Unknown

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (focus group): Participants attend a focus group session and review printed copies of planned posts for the to-be-developed Facebook intervention over 90 minutes to 2 hours.
  Interventions: Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This research trial collects feedbacks from indoor tanning bed users via focus group for the development of social media-delivered intervention. Conducting a focus group with people using indoor tanning bed and having access to Facebook may help doctors to better understand people's perspective and thoughts about the various Facebook messages.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To elicit feedback from young adult women who use indoor tanning beds on preliminary intervention content.

OUTLINE:

Participants attend a focus group session and review printed copies of planned posts for the to-be-developed Facebook intervention over 90 minutes to 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Use of an indoor tanning bed at least 10 times in the past 12 months
* At least daily use of Facebook

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Facebook users use of an indoor tanning bed at least 10 times in the past 12 months
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
Participants feedback | Up to 2 years
  Focus group questions will elicit descriptions of general interest. Participants will also rate various posts on the hand-out sheets included in the script.
Participants feedback | Up to 2 years
  Focus group questions will elicit descriptions of posts, and as well as suggestions for improving existing posts or creating new ones. Participants will also rate various posts on the hand-out sheets included in the script.
Participants feedback | Up to 2 years
  Focus group questions will elicit descriptions of general interest of topics. Participants will also rate various posts on the hand-out sheets included in the script.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No